CLINICAL TRIAL: NCT03730402
Title: Laparoscopic Assisted Plane Block (LAPB) Trial: Bupivacaine Versus Liposomal Bupivacaine Versus Standard Local Anesthesia for Post-operative Analgesia
Brief Title: Laparoscopic Assisted Plane Block (LAPB) Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There were not enough attendings/residents working on the study throughout the COVID-19 pandemic in order to enroll the number of patients required to meet statistical significance.
Sponsor: Santa Barbara Cottage Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18-66mr
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Opioid Use
Keywords: post-operative analgesia
MeSH Terms: interventions — Bupivacaine; Injections; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: prospective randomized control trial
Who Masked: Participant
Masking Description: single-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- bupivacaine block (Active Comparator): laparoscopic assisted plane block of standardized dose of bupivacaine plain
  Interventions: Drug: Bupivacaine
- liposomal bupivacaine block (Exparel 266 milligram Per 20 ML) (Active Comparator): laparoscopic assisted plane block of standardized dose of bupivacaine plain
  Interventions: Drug: Exparel 266 milligram Per 20 ML Injection
- saline block (Placebo Comparator): laparoscopic assisted plane block with placebo saline injection
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — utilizing local anesthetic to perform a regional block under laparoscopic guidance
  Other Names: Marcaine
  Arms: bupivacaine block
Drug: Exparel 266 milligram Per 20 ML Injection — utilizing local anesthetic to perform a regional block under laparoscopic guidance
  Other Names: Exparel, liposomal bupivacaine
  Arms: liposomal bupivacaine block (Exparel 266 milligram Per 20 ML)
Drug: Saline — placebo injection of saline
  Other Names: Injectable Saline
  Arms: saline block

SUMMARY:
This study attempts to demonstrate improvement in analgesia in a more diverse laparoscopic surgery group with the use of laparoscopic assisted transversus abdominis plane blocks. The investigators will compare bupivacaine (treatment arm 1) versus liposomal bupivacaine (treatment arm 2) versus port site injection of local anesthesia with injection of saline placebo (control). The hypothesis is that liposomal bupivacaine will result in improved analgesia when compared to bupivacaine LAPB and control. The investigators further hypothesize that bupivacaine LAPB will be more effective than the control.

DETAILED DESCRIPTION:
Patients will either be pre-screened prior to their pre-operative appointment for eligibility, or screening will occur on the day of surgery. Informed Consent will be obtained from amenable, eligible patients prior to their operation by a member of the research team. A study number will be assigned, and the patient will be randomized to a treatment group. The patients will not be aware to which treatment group they have been randomized.

After consent is obtained and randomization has been completed, the operating room registered nurse will calculate maximum dose of allowable bupivacaine per patient based on body weight. Anesthesia will provide the intravenous lidocaine bolus on induction to all patients without a contraindication to the medication. The port placement will occur using a needle to raise skin/preperitoneal wheal*. Up to 20cc of 1% lidocaine/epinephrine will be divided among all ports and stab incisions. At end of case, no further skin or port-specific preperitoneal anesthetic will be injected unless a skin incision was extended.

For patients randomized to port site injection (Control): 60 cc of sterile, preservative-free, injectable saline will be given as a placebo per the protocol in item 6.

For patients randomized to bupivacaine plain LAPB (Treatment Arm 1): The maximum weight-based dose of plain bupivacaine will be diluted with sterile, injectable, preservative-free saline to a total of 60cc with a maximum of 250mg bupivacaine (regardless of weight) and loaded into a 30cc syringe with a 22g spinal needle (one 30cc syringe used for each side).

For patients randomized to liposomal bupivacaine LAPB (Treatment Arm 2): The maximum dose for adult patients is 266mg (20mL) of liposomal bupivacaine. This will be diluted with 40cc of preservative-free normal saline for injection, per manufacturer recommendations. The solution will then be loaded into a 30cc syringe with a 22g spinal needle and injected in the same fashion as the bupivacaine plain LAPB.

Data collection will include total doses of IV and skin and block anesthetic used, patient weight, number and size of ports, if fascial closure of port site was conducted, and post-operative narcotic medication used up to 48 hours with timing and doses marked, and use of any pain adjuncts (nonsteroidal anti-inflammatory drugs [NSAIDs], acetaminophen, gabapentin, tricyclic antidepressants [TCA], pregabalin, clonidine, etc.) although doses of these medications are not to be recorded.

Provision of home narcotic prescription will be based on a standardized protocol developed by Dartmouth. Based on the past 24 hours of pain medication usage, patients will receive either 15 or 30 tablets of hydrocodone/acetaminophen 5/325mg (or liquid equivalent for bariatric patients). Use of narcotic medications at home will be evaluated at 1 week post-procedure by a member of the research team through a phone survey.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years old
* Patients undergoing non-emergent laparoscopic surgery with planned or continued admission for at least 1 night
* Patients who receive fully laparoscopic procedures including ports up to 15mm, and any blunt dilation of port fascia or sharp extension of skin incisions for specimen extraction.

Exclusion Criteria:

* Patients under 18 or over 80 years old
* Patients who are pregnant
* Patients who are unable to consent themselves
* Patients who undergo an appendectomy for acute appendicitis
* Patients who undergo emergent surgery
* Patients who are converted to open procedure
* Patients who receive concurrent neuraxial anesthesia (spinal, epidural, or indwelling pain pumps)
* Patients who receive concurrent local anesthetic drips planned during or administered immediately after surgery
* Patients who have a contraindication to local anesthetics (e.g. verified allergy, severe hepatic dysfunction)
* Patients who use chronic narcotics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Narcotic Usage | 24 hours
  post-operative narcotic usage expressed in morphine equivalents

SECONDARY OUTCOMES:
Narcotic Usage | 7 days
  post-operative narcotic usage expressed in morphine equivalents
Pain Scores | 24 hours
  Visual Analog Score for pain (1-10)
Post-Operative Nausea | 24 hours
  Post-operative nausea will be quantified through chart review by recording the amount of anti-emetic medication administered in the 24 hour period the patient is admitted post-operatively. This will allow objective quantification of nausea in the immediate post-operative period for analysis.
Post-operative emesis | 24 hours
  Emesis is recorded as part of the standard intake/output medical charting, and the number of episodes of emesis will be quantified from chart review. This will be analyzed between groups to determine if the intervention has an impact on the number of episodes of post-operative emesis.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Zerey, MD, Principal Investigator — Cottage Hospital, Sansum Clinic
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No